CLINICAL TRIAL: NCT01497574
Title: A Single-centre, Randomised, Double-blind, Cross-over Trial Comparing the Within-subject Variability of the Pharmacokinetic Profiles of Insulin Detemir and Insulin Glargine in Children and Adolescents With Type 1 Diabetes
Brief Title: Within-subject Variability of Insulin Detemir in Children and Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN304-1633; 2004-001692-19 (EudraCT Number)
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin detemir (Experimental)
  Interventions: Drug: insulin detemir; Drug: insulin glargine
- Insulin glargine (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin glargine

INTERVENTIONS:
Drug: insulin detemir — On two dosing visits, 0.4 U/kg insulin detemir will be administered followed by 0.4 U/kg insulin glargine after a 24 hours' interval and repeated in opposite order at next dosing visit. Administrated subcutaneously (s.c., under the skin)
Drug: insulin glargine — On two dosing visits, 0.4 U/kg insulin glargine will be administered followed by 0.4 U/kg insulin detemir after a 24 hours' interval and repeated in opposite order at next dosing visit. Administrated subcutaneously (s.c., under the skin)

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the within-subject variability of the pharmacokinetic profiles of insulin detemir and insulin glargine in children and adolescents with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Body mass index (BMI) for children (6 to 12 years): 15-20 kg/m^2 (both inclusive)
* Body mass index (BMI) for adolescents (13 to 17 years): 18-25 kg/m^2 (both inclusive)
* HbA1c (glycosylated haemoglobin) below 11.0% according to central laboratory results
* Current treatment with insulin at least twice daily

Exclusion Criteria:

* Any significant disease such as endocrine, hepatic, renal, cardiac, neurological, malignant, or pancreatic disease other than diabetes
* Receipt of any investigational product within the last four weeks
* Known or suspected allergy to trial products or related products

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2005-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Area under the insulin concentration curve (AUC)

SECONDARY OUTCOMES:
Maximum insulin concentration (Cmax)
Time to maximum insulin concentration (tmax)
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Hanover, Germany

REFERENCES:
- [Result] Danne T, Datz N, Endahl L, Haahr H, Nestoris C, Westergaard L, Fjording MS, Kordonouri O. Insulin detemir is characterized by a more reproducible pharmacokinetic profile than insulin glargine in children and adolescents with type 1 diabetes: results from a randomized, double-blind, controlled trial. Pediatr Diabetes. 2008 Dec;9(6):554-60. doi: 10.1111/j.1399-5448.2008.00443.x. Epub 2008 Aug 27. PMID 18761644
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com